CLINICAL TRIAL: NCT05569278
Title: A Phase 1 Single Centre, Single Ascending Dose Safety Study of GEH200486 in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of GEH200486 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GE-227-001; 2021-005791-19 (EudraCT Number)
Record Dates: First submitted 2022-08-17; First posted 2022-10-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GEH200486 Cohort 1 (Experimental): Participants will receive 0.05 mmol/kg of GE200486 0.5 M injection
  Interventions: Drug: GE200486 0.5M Injection
- GEH200486 Cohort 2 (Experimental): Participants will receive 0.1 mmol/kg of GE200486 0.5 M injection
  Interventions: Drug: GE200486 0.5M Injection
- GEH200486 Cohort 3 (Experimental): Participants will receive 0.2 mmol/kg of GE200486 0.5 M injection
  Interventions: Drug: GE200486 0.5M Injection
- GEH200486 Cohort 4 (Experimental): Participants will receive 0.3 mmol/kg of GE200486 0.5 M injection
  Interventions: Drug: GE200486 0.5M Injection

INTERVENTIONS:
Drug: GE200486 0.5M Injection — Single administration by intravenous (IV) hand injection without dilution, followed by a 5mL saline flush

SUMMARY:
This is a single center, prospective, dose escalation study (4 different dose levels) for a novel magnetic resonance imaging (MRI) contrast agent, in male and female healthy volunteers . The study is primarily designed to collect safety data. In addition, researchers want to learn more about how the novel contrast agent, GEH200486 circulates and is eliminated from the body (pharmacokinetics) after injection in healthy volunteers. Up to 24 healthy volunteers will be enrolled and will each receive a single administration of one of the 4 doses of GEH200486. Each healthy volunteer will stay at the clinical unit for the first 24 hours post injection and return for up to 3 follow-up visits with 1 additional follow-up phone call.

Dose escalation from one dose group to the next dose group will be sequential and only be allowed if the clinical safety of all healthy volunteers from the tested dose group is acceptable, as assessed by an independent safety committee, members of GEHC team and the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 18 to 55 years of age
* The subject has no currently active significant medical illness or history of chronic medical illness.
* The subject has no clinically significant deviation from normal ranges in physical examination, ECG, and clinical laboratory parameters.
* The subject has read, signed, and dated an informed consent form (ICF) prior to any study procedures being performed, and is willing to allow the study Investigator to make the subject's medical records available to GE Healthcare
* The subject is able and willing to comply with all study procedures as described in the protocol.
* Female subjects: The subject is a female who is either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (amenorrhoea duration of at least 12 consecutive months), or non- lactating, or if of childbearing potential the results of a urine human chorionic gonadotropin pregnancy test, performed at screening and on the day of dosing, prior to administration (with the result known before investigational medicinal product [IMP] administration), must be negative. Women of childbearing potential must use adequate contraception from screening until 30 days after administration of IMP. Such methods include: hormonal contraception including oral contraceptives; intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion; vasectomised partner; sexual abstinence.
* Male subjects: The subject is a male who is either surgically sterile or males who are sexually active with a partner of childbearing potential must use adequate contraception from screening until 30 days after administration of IMP. Such methods include: vasectomy; sexual abstinence. Male subjects must agree not to donate sperm from screening through 30 days after administration of IMP

Exclusion Criteria:

* Subjects who are unable to undergo any of the study procedures.
* Subjects with any significant currently active or chronic medical illness (e.g., cardiovascular disease, renal impairment, hepatic dysfunction, Parkinson's disease) or recent significant trauma (e.g., motor vehicle accident) or any condition that may have disrupted and/or increased permeability of the blood-brain barrier.
* Subjects with any major surgery within 4 weeks prior to enrolment or planned within 2 weeks after completion of the study.
* Subjects who have a positive urine screen for alcohol and/or recreational drugs at screening or before dosing.
* Subjects who are taking prescribed medication (other than contraception) within 2 weeks prior to enrolment or anticipate using prescribed medication (other than oral contraception) during the enrolment period through study follow-up. Limited use of non- prescription medications which in the Investigator's opinion will not affect subject safety or the overall results of the study may be permitted (e.g., acetaminophen/paracetamol) on a case-by-case basis following approval by the Sponsor.
* Subjects who have undergone a contrast-enhanced (CE) imaging procedure (CE-MRI, CE computed tomography [CT]) during the 30 days prior to dosing.
* Subjects who are taking any concomitant medications or dietary supplements that are known to increase blood levels of Mn, Zn, copper (Cu), or iron (Fe) for the duration of the study.
* Subjects who have serious allergic history or known or suspected allergy to the study drug GEH200486 0.5 M Injection or study drug ingredients.
* Subjects who present with any clinically active, serious, life-threatening disease, medical or psychiatric condition, known abuse or misuse of prescription or non-prescription drugs and subjects whom the Investigator judges to be unsuitable for participation in the study for any reason.
* Subjects with previous (within 30 days before administration of IMP or within 5 half-lives of the investigational treatment of the previous study, whichever is longer) or concomitant participation in another clinical study with IMP(s).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Collection of occurrence of IMP-related SAEs | After administration of IMP until 72 hours post dose (up to 17 days post dose)
Collection of TEAEs | After administration of IMP until 72 hours post dose (up to 17 days post dose)
Collection of AEs | After administration of IMP until 72 hours post dose (up to 17 days post dose)
Injection site monitoring findings at pre-specified time points. | Continuous monitoring from IMP injection up to 24 hours
Change from baseline in the results of serum biochemistry test results at pre-specified time points. | Baseline, 1 hour, 4 hours, 24 hours, 48 hours and 72 hours post IMP administration
  In this context, baseline is defined as the pre-treatment assessment at the screening visit. The occurrence of post injection values outside of normal limits and changes from baseline will be summarized.
Change from baseline in the results of urinalysis at pre-specified time points. | Baseline, 48 hours and 72 hours post IMP administration
  In this context, baseline is defined as the pre-treatment assessment at the screening visit. The occurrence of post injection values outside of normal limits and changes from baseline will be summarized.
Change from baseline in the results of haematology at pre-specified time points. | Baseline, 1 hour, 4 hours, 24 hours, 48 hours and 72 hours post IMP administration
  In this context, baseline is defined as the pre-treatment assessment at the screening visit. The occurrence of post injection values outside of normal limits and changes from baseline will be summarized.
Measure of blood pressure in mmHg at pre-specified time points | Baseline, 10 minutes, 30 minutes, 1 hour, 4 hours, 24 hours, 48 hours and 72 hours post IMP administration
Measure of body temperature as degree C at pre-specified time points | Baseline, 10 minutes, 30 minutes, 1 hour, 4 hours, 24 hours, 48 hours and 72 hours post IMP administration
Measure of heart rate as bpm at pre-specified time points | Baseline, 10 minutes, 30 minutes, 1 hour, 4 hours, 24 hours, 48 hours and 72 hours post IMP administration.
Measure of respiratory rate per min at pre-specified time points | Baseline, 10 minutes, 30 minutes, 1 hour, 4 hours, 24 hours, 48 hours and 72 hours post IMP administration

SECONDARY OUTCOMES:
Pharmacokinetic assessment | pre-dose to 24 hours
  AUC0-t Area under the concentration versus time curve (AUC) from time zero to the last measurable concentration, calculated using the linear up/log down trapezoidal rule.
Change from baseline in the results of ECG examinations (PR interval, QTc, QRS and RR interval) at pre-specified time points. | Baseline (prior to IMP administration) up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Francois Tranquart, MD, PhD, Study Director — GE Healthcare
Locations (1):
- Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No